CLINICAL TRIAL: NCT03949322
Title: Physical Activity, Cancer and Cognitive Function Disorders : Effects of an Adapted Physical Activity Program on Impaired Cognitive Function in the Management of Cancer
Brief Title: Cancer Related Cognitive Impairment
Acronym: APACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: University of Poitiers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-N-2018-21
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Patients Treated for Cancer
Keywords: physical activity; cancer Related Cognitive Impairment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Physical Activity Program (Experimental): Patients in the experimental group take part in a program of Adapted Physical Activity lasting 6 weeks, with 2 sessions per week.
  Interventions: Behavioral: Adapted Physical Activity Program

INTERVENTIONS:
Behavioral: Adapted Physical Activity Program — The sessions in this program are similar to the adapted physical activity sessions already offered by sports therapy practitioners. This is an aerobic exercise session, with Nordic walking, and a combined session of muscle building and breathing exercises.

SUMMARY:
Various recent scientific data testify to the cognitive deficiencies of cancer patients, called Cancer-Related Cognitive Impairments (CRCI) (Noal, Daireaux & Joly, 2010). At the same time, regular physical activity (aerobic, muscle building, and yoga) has been shown to decrease CRCIs, although commonly used cognitive measures are self-reported (Zimmer et al., 2016). The investigators will develop an interventional study using objective measures of cognition to confirm the cause-and-effect relationship, and specify the orientation of the cognitive effects of the adapted physical activities. The main and original objective will be to determine if the cognitive functions most affected by CRCI (episodic memory, inhibition, treatment speed) can be optimized in patients undergoing treatment.

DETAILED DESCRIPTION:
1. Inclusion procedure and saving selection failures Participation in this study will be offered to patients during their care in day hospital (= inclusion visit).

   Any patient giving express consent to participation and meeting the criteria for inclusion and non-inclusion will then be included in the study.

   Each patient will then be identified by his or her initials as a patient number in the study, directly on the basis of collecting the data from the study.
2. Study progress for patients Data collection takes place over two different periods. Each period lasts 12 weeks. The Adapted Physical Activity (APA) program is 8 weeks old.

The first period will run from mid-January to early April (first cohort) to collect data from the first patients in the experimental group.

The second period will be from mid-February to the end of April. During this one, it will be necessary to collect the data of the last patients of the experimental group (second cohort) The first two weeks of each period (weeks 1 and 2, weeks 4 and 5) are dedicated to recruiting patients.

During the pre-test session, carried out week 3 for the first cohort and weeks 6 for the second, the patients will carry out different tests and questionnaires: General Information Questionnaires, Education, MoCA (Montreal Cognitive Assessment), GPAQ (Global Physical Activity Questionnaire), Stroop test, test of MEM3 (Echelle Clinique de Mémoire), letter comparison test, HADS (Hospital and Anxiety Depression Scale), and the MFI (Multidimensional Fatigue Inventory). Patients should also wear an actimeter for one week from the day of recruitment.

Patients then take part in a program of Adapted Physical Activity lasting 8 weeks, with 2 sessions per week. The sessions of this program are similar to the APA sessions already offered by sports therapy practitioners. This is an aerobic exercise session, with Nordic walking, and a combined session of muscle building and breathing-based exercises.

In the post-test session, which was conducted week 12 for the first cohort and week 15 for the second, some questionnaires and tests are again administered: GPAQ, Stroop test, MEM3 test, letter comparison test, HADS and the MFI. Patients should also wear an actimeter the week before the day of the post-test.

The forecast schedule may be slightly modified depending on unforeseen circumstances and constraints that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female> or = 18 years old
2. Any patient being treated for a cancerous condition and managed by adjuvant chemotherapy.
3. Any type of cancer
4. Beneficiary of a social protection scheme
5. Having as mother tongue the French language
6. Patient information and obtaining express consent

Exclusion Criteria:

1. Protected subjects known as vulnerable (major under legal protection, adults unable to express their consent, subject admitted to a health and social institution).
2. Minor subjects
3. Pregnant women, likely to be pregnant or breastfeeding
4. Subjects with sensory disabilities affecting vision or hearing
5. Neurological or psychiatric antecedents
6. Persons deprived of liberty or guardianship (including trusteeship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Effect of an APA program on cognitive functions (inhibition) | 8 weeks
  For inhibition, effect of APA program on cognitive functions is evaluated with Stroop task.
Effect of an APA program on cognitive functions (speed function of information processing) | 8 weeks
  For speed function of information processing, effect of APA program on cognitive functions is evaluated with XO letters comparison test. During the XO letters comparison test, the participants will have to check the maximum number of identical or different boxes according to the combination of the two letters presented (XO, OX, XX or OO) in 30 seconds.
Effect of an APA program on cognitive functions (Episodic Memory Function) | 8 weeks
  For Episodic Memory Function, effect of APA program on cognitive functions is evaluated with MEM III test.

SECONDARY OUTCOMES:
To determine if the APA program modifies PA (Physical Activity) patterns in daily life | 8 weeks
  Evaluated with Global Physical Activity Questionnaire
To determine if the APA program modifies PA (Physical Activity) patterns in daily life | 8 weeks
  Evaluated with Actimeter
Determine which PA pattern is the best predictor of cognitive performance improvement following the APA program, , by controlling the effect of cognitive risk factors. | 8 weeks
  Level of overall cognitive abilities: Montreal Cognitive Assessment (MOCA)
Determine which PA pattern is the best predictor of cognitive performance improvement following the APA program, , by controlling the effect of cognitive risk factors. | 8 weeks
  Level of education: questionnaire measuring the number of years of study
Determine which PA pattern is the best predictor of cognitive performance improvement following the APA program, , by controlling the effect of cognitive risk factors. | 8 weeks
  Level of Anxiety and Depression: Hospital and Anxiety Depression Scale (HADS).
Determine which PA pattern is the best predictor of cognitive performance improvement following the APA program, , by controlling the effect of cognitive risk factors. | 8 weeks
  Fatigue level: Multidimensional Fatigue Inventor (MFI)

CONTACTS AND LOCATIONS:
Overall Officials: BOIFFARD Florence, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, France